Augmented Macular Pigment Supplement and Pericentral Visual Function: A Randomized Controlled Trial

NCT #: NCT04676126

Date: 28 April 2021

## Subject Consent to Take Part in a Study of

## VISUALL-3: A VISUAL ACUITY VALIDATION STUDY University of the Incarnate Word Baptist Medical Center Glaucoma Service

**Authorized Study Personnel:** William Sponsel, MD, Principal-Investigator

Baptist Medical Center Glaucoma Service

210-223-9292

sponsel@earthlink.net

Grant Slagle, DO, Co-Investigator Research Fellow, Sponsel Foundation

561-789-3640

slaglegrant@gmail.com

**Key Information:** Your consent is being sought for a research study. The purpose of the research is to validate a new device for vision testing. If you agree to participate in this study, the project will involve:

- Taking an oral supplement + eye drop (or placebo) that contains nutrients that we think might improve your vision
- 4 visits are required
- Each visit will be approximately 2 hours long and will involve testing:
  - Contrast Sensitivity
  - Density of macular pigments
  - Skin macular pigment levels (Veggie Meter)
  - At your first and final visit you will do a visual field test (FDT)
- There are minimal risks associated with this study
- You will receive compensation in the form of gift cards for your participation in this study
- Your participation is voluntary and you may decide not to participate at any time

**Invitation:** You are invited to volunteer as one of 30 subjects in the research project named above. The information in this form is meant to help you decide whether or not to participate. If you have any questions, please ask.

Why are you being asked to be in this research study? You are being asked to be in this study because you are an adult with glaucoma with good eye pressure control but you still appear to be losing vision on the visual field test.

What is the reason for doing this research study? The purpose of this study is to see if there is any improvement in visual function or measurements of macular pigments in your skin and eye. Macular pigments are nutrients that are important for protecting your eye from harmful light. The supplement we are asking you to take contains these nutrients.

What will be done during this research study? We will randomly assign you to receive Lumega-Z + dorzolamide (supplement with macular pigments) or a placebo (a similar drink without active ingredients) and then test to see how taking the supplement or placebo affects nutrient levels in your skin and eye. We will also test how well you can identify contrast, and how your visual field may be affected.

This study is not part of your health care.

**How will my data/samples/images be used?** Your specific data could be used for future research studies. You are given the option to choose whether you will allow your deidentified data to be stored indefinitely for further analysis or other relevant research studies.

## Will I be notified if my data result(s) in an unexpected finding?

When specific data are collected and analyzed, there is a chance of finding something unexpected. There may be benefits to learning such results (such as early detection and treatment of a medical condition), but there are risks as well (such as feeling worried about a finding for which no treatment is needed).

In this study, you will be informed of any unexpected findings of possible clinical significance that may be discovered during review of results from your data. The results from the data we collect in this research are not the same as what you would receive as part of your health care. The data will be reviewed by a physician who normally reads such results and if there are any unexpected findings and we will provide you with this information so that you may discuss it with your personal physician. If you believe you are having symptoms that may require care prior to receiving any information from this study, you should contact your personal physician.

What are the possible risks of being in this study? There are minimal risks to you from being in this research study.

-Minor pain or discomfort: The eye drop may cause some minor discomfort on the eye. It is usually not severe enough to warrant stopping the drop. Please let us know if the drop causes severe burning or pain.

-COVID-19: we exceed CDC recommendations in order to ensure you are safe while you are at the office

What are the possible benefits to you? It is possible that the supplement you take will cause a small improvement in vision, but it is also possible that nothing will happen.

What are the possible benefits to other people? The potential benefits of taking a supplement like Lumega-Z are not yet fully known. If we find that it is beneficial for glaucoma patients, many patients with glaucoma may start taking the medication and also benefit.

What are the alternatives to being in this research study? Instead of being in this research study you can choose not to participate.

What will being in this research study cost you? There is no cost to you to be in this research study.

**Will you be compensated for being in this research study?** You will be awarded a gift card at the end of each visit of the following amounts:

Visit 1: \$25

Visit 2: \$25

Visit 3: \$25

Visit 4: \$100

**How will information about you be protected?** Everything we learn about you in the study will be confidential. The only persons who will have access to your research records are the study personnel, the

Institutional Review Board (IRB), and any other person, agency, or sponsor as required by law. If we publish with results of the study, you will not be identified in any way.

What will happen if you decide not to be in this research study or decide to stop participating once you start? You can decide not to be in this research study, or you can stop being in this research study at any time, for any reason. Deciding not to be in this research study or deciding to withdraw will not affect your relationship with the investigator or with the University of the Incarnate Word or Baptist Medical Center Glaucoma Service. You will not lose any benefits to which you are entitled.

What should you do if you have a problem or question during this research study? If you have a problem as a direct result of being in this study, you should immediately contact one of the people listed at the beginning of this consent form.

If you have any questions now, feel free to ask us. If you have additional questions about your rights or wish to report a problem that may be related to the study, please contact the University of the Incarnate Word Institutional Review Board office at 210-805-3036 or 210-805-3565.

| Consent for future use of data: Initial one of the following to indicate your choice: | |
|---|---|
| I give permission for my deidentified data to be relevant research studies. I understand that no additiounderstand that my deidentified data can be stored inc | |
| I give my permission for my data to be used for for any future use beyond the scope of this research s within 2 years after completion of this study. | this research study only. I do not give permission tudy. I understand that my data will be destroyed |
| Consent Your signature indicates that you (1) consent to take part in this research study, (2) that you have read and understand the information given above, and (3) that the information above was explained to you, and you have been given the chance to discuss it and ask questions. You will be given a copy of this consent form to keep. | |
| Name of Participant | |
| Signature of Participant | Date |
| Name of Principal Investigator/Designee | |

Date

Signature of Principal Investigator/Designee